CLINICAL TRIAL: NCT00003962
Title: Dose Finding Study of Toxicity and Immunomodulatory Effects of Interleukin-2 Following Allogeneic Bone Marrow Transplantation in Patients at High Risk for Relapse
Brief Title: Interleukin-2 Following Bone Marrow Transplantation in Treating Patients With Hematologic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: J9825 CDR0000067162; P01CA015396 (NIH); JHOC-98040902; JHOC-J9825; NCI-H99-0033
Record Dates: First submitted 1999-11-01; First posted 2004-08-27 (Estimated); Last update posted 2014-05-02 (Estimated); Status verified 2014-05

CONDITIONS: Leukemia; Lymphoma; Multiple Myeloma and Plasma Cell Neoplasm
Keywords: recurrent childhood acute lymphoblastic leukemia; recurrent adult Hodgkin lymphoma; refractory multiple myeloma; stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma; recurrent childhood lymphoblastic lymphoma; recurrent childhood acute myeloid leukemia; recurrent adult acute myeloid leukemia; recurrent adult acute lymphoblastic leukemia; recurrent/refractory childhood Hodgkin lymphoma; chronic myelomonocytic leukemia; acute undifferentiated leukemia; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult T-cell leukemia/lymphoma; secondary acute myeloid leukemia; AIDS-related peripheral/systemic lymphoma; recurrent childhood small noncleaved cell lymphoma; recurrent childhood large cell lymphoma; recurrent mantle cell lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma
MeSH Terms: conditions — Leukemia; Lymphoma; Multiple Myeloma; Neoplasms, Plasma Cell; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Hodgkin Disease; Leukemia, Myeloid, Acute; Recurrence; Leukemia, Myelomonocytic, Chronic; Leukemia, Biphenotypic, Acute; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Burkitt Lymphoma; Dendritic Cell Sarcoma, Interdigitating; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — aldesleukin

INTERVENTIONS:
Biological: aldesleukin

SUMMARY:
RATIONALE: Interleukin-2 may stimulate a person's white blood cells to kill cancer cells.

PURPOSE: Phase I trial to study the effectiveness of interleukin-2 following bone marrow transplantation in treating patients who have hematologic cancer at risk of relapse.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the toxicity and maximum tolerated dose of interleukin-2 following allogeneic T-cell depleted bone marrow transplant in patients with hematologic malignancies at high risk of relapse. II. Determine the optimal dose of interleukin-2 in this regimen which will result in maximal natural killer cell and lymphokine activated killer cell activity in vitro.

OUTLINE: This is a dose escalation study. Patients receive CD34+ stem cell augmented donor bone marrow on day 0 on another protocol. Patients then receive interleukin-2 (IL-2) subcutaneously on day 30. Treatment continues for 12 weeks in the absence of dose limiting toxicity. Cohorts of 4 patients receive escalating doses of IL-2 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose prior to that which causes at least grade 3 toxicity.

PROJECTED ACCRUAL: A total of 18-24 patients will be accrued for this study within 12-18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Any of the following diagnoses eligible: Acute myelogenous leukemia beyond first complete remission Acute lymphoblastic leukemia Chemotherapy resistant non-Hodgkin's lymphoma Chemotherapy resistant Hodgkin's disease Multiple myeloma Primary refractory acute leukemia Secondary leukemia Chronic myelomonocytic leukemia No chronic myelogenous leukemia, aplastic anemia, or myelofibrosis HLA identical related donor required

PATIENT CHARACTERISTICS: Age: 0.5 to 65 Performance status: ECOG 0-2 Life expectancy: Not specified Hematopoietic: See Disease Characterisitics Hepatic: Bilirubin less than 2.5 mg/dL (unless Gilbert's syndrome present) Renal: Creatinine no greater than 2 mg/dL Cardiovascular: No active congestive heart failure, arrhythmia, or angina pectoris No myocardial infarction within past 12 months Pulmonary: No requirement for oxygen Other: Afebrile for greater than 48 hours No active, serious infection (e.g., sepsis, mucormycosis, or uncontrolled aspergillosis) No debilitating medical or psychiatric illness that would preclude compliance Not pregnant Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: No prior bone marrow transplant Chemotherapy: See Disease Characteristics Endocrine therapy: No concurrent corticosteroids Radiotherapy: Not specified Surgery: Not specified

Max Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1998-04; Primary Completion 2000-06 (Actual); Study Completion 2000-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul V. O'Donnell, MD, PhD, Study Chair — Fred Hutchinson Cancer Center
Locations (1):
- Johns Hopkins Oncology Center, Baltimore, Maryland, United States